CLINICAL TRIAL: NCT02747238
Title: Does Ultrasound-guided CSE Technique Improve Midline Placement of Epidural Needle Thereby Helping Junior Residents With Correct Placement of the Catheter Compared to the Placement Using With Anatomical Landmarks?
Brief Title: Does Ultrasound Help Junior Anesthesia Residents With Placement of Labor Analgesia in Pregnant Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Barbara S Orlando, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 15-1180
Record Dates: First submitted 2015-06-03; First posted 2016-04-21 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy
Keywords: Pregnancy; Epidural; Labor
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ultrasound (Active Comparator): Woman requests epidural for pain relief Ultrasound guided CSE placed Continuous epidural infusion started
  Interventions: Device: Ultrasound; Procedure: Epidural infusion
- No ultrasound (Active Comparator): Palpation of anatomical landmarks Woman requests epidural for pain relief CSE placed using palpation of anatomical landmarks Continuous epidural infusion started
  Interventions: Procedure: No ultrasound; Procedure: Epidural infusion

INTERVENTIONS:
Device: Ultrasound — The ultrasound imaging of the lumbar spine in different scanning planes facilitates the identification of the landmarks necessary for appropriate epidural space location in pregnant patients. There are two acoustic windows that are effective for lumbar spine sonographic assessment: one seen on the transverse approach, and the other seen on the longitudinal paramedian approach. The ultrasound single-screen method using the transverse approach of the lumbar spine provides reliable information regarding the landmarks required for labor epidurals. The correct interspace and midline position are identified for correct placement of the CSE analgesia.
  Arms: Ultrasound
Procedure: No ultrasound — Palpation of anatomical landmarks is used for placement of labor analgesia
  Arms: No ultrasound
Procedure: Epidural infusion — An epidural infusion will be started in both groups, regarding of the technique used for placement, and the same solution of Bupivacaine 0.0625% with 2mcg fentanyl/cc will be used in both groups

SUMMARY:
The investigators believe that ultrasound guided CSE technique will help junior resident rotating for the first time on the labor and delivery floor to place more accurately the epidural needle in the midline position as compared to placing the epidural needle via palpation of anatomical landmarks. This will result in increased ability to place the spinal component with positive cerebral spinal fluid (CSF) in the spinal needle, correct midline placement of the epidural catheter, and increase the likelihood of adequate symmetrical labor analgesia/anesthesia.

DETAILED DESCRIPTION:
Epidurals provide superior labor analgesia and anesthesia. Unfortunately, failure of epidural anesthesia and analgesia is a frequent clinical problem. In a heterogeneous cohort of 2,140 surgical patients, a failure rate of 27% for lumbar epidural was described. However, the definition of a failed epidural is broad. Different definitions include insufficient analgesia to catheter dislodgement to conversion to general anesthesia. Epidural analgesia failures may result from technical difficulties, insufficiencies or overdosing of local anesthetics, epidural septum or midline adhesions, and placement of the epidural catheter through an intervertebral foramen or into the anterior epidural space. In an imaging study of failed epidurals, incorrect catheter placement accounted for half of the failures, while the remaining patients experienced suboptimal analgesia through a correctly positioned catheter.

The incidence of overall failure was lower in patients receiving combined spinal-epidural (CSE) catheters versus epidural analgesia. In one study, the CSE technique provided decreased failure rates for labor analgesia and comparable or decreased failure rates for surgical anesthesia, when compared with reported failure rates for epidural anesthesia. It is believed that positive CSF flow in the spinal needle confirms correct epidural needle placement in the epidural space and also confirms the epidural needle to be in the midline position. Placement of the epidural needle in the midline position will minimize the incorrect placement of the catheter to one side, providing a symmetrical analgesia versus unilateral analgesia.

However, the practice of CSE and epidural catheter placement relies on the palpation of anatomical landmarks that are not always easy to feel. Therefore, the epidural needle maybe placed "off midline" despite positive loss of resistance (LOR) that causes negative CSF flow in the spinal needle and an incorrectly placed catheter. As a result, the incorrect catheter placement will result in a "failed" or suboptimal epidural analgesia.

Ultrasound has recently been utilized to facilitate lumbar epidurals and spinals. The US imaging of the lumbar spine in different scanning planes facilitates the identification of the landmarks necessary for appropriate epidural space location in pregnant patients. There are two acoustic windows that are effective for lumbar spine sonographic assessment: one seen on the transverse approach, and the other seen on the longitudinal paramedian approach. The ultrasound single-screen method using the transverse approach of the lumbar spine provides reliable information regarding the landmarks required for labor epidurals. The correct interspace and midline position are identified for correct placement of the CSE analgesia.

A previous study done by the research team, comparing "blind" vs US guidance technique. It did not show any significant difference in term of success rate or complications with either technique. However, the study was done by 4 trained physicians with lot of practice. At this level of training, the investigators did not observe any technique improvement with US. Which is why the investigators thought might have more success in showing an improvement in technique, with junior residents rotating for the first time on the floor. The idea is to see if there is any difference in their learning curve using the US versus the "blind" technique. Each resident will be their own control.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Term (>37 weeks gestation)
* Vertex presentation
* Singleton gestation
* Ability to provide informed consent
* Request for analgesia for labor pain
* Maternal age 18 years or greater

Exclusion Criteria:

* Multiparous
* Preterm (< 37 weeks gestation)
* Presentation other than vertex (breech, transverse)
* Active drug/alcohol dependence
* Previous spinal surgeries
* Known spinal deformities

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Orlando, MD, Principal Investigator — Mount-Sinai Roosevelt Hospital
Locations (1):
- Mount-Sinai Roosevelt Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound: Patients that had Ultrasound guided CSE placed
  Ultrasound: The ultrasound imaging of the lumbar spine in different scanning planes facilitates the identification of the landmarks necessary for appropriate epidural space location in pregnant patients. There are two acoustic windows that are effective for lumbar spine sonographic assessment: one seen on the transverse approach, and the other seen on the longitudinal paramedian approach. The ultrasound single-screen method using the transverse approach of the lumbar spine provides reliable information regarding the landmarks required for labor epidurals. The correct interspace and midline position are identified for correct placement of the CSE analgesia.
  Epidural infusion: An epidural infusion will be started in both groups, regarding of the technique used for placement, and the same solution of Bupivacaine 0.0625% with 2mcg fentanyl/cc will be used in both groups
- No Ultrasound: Patients that had CSE placed using palpation of anatomical landmarks
  No ultrasound: Palpation of anatomical landmarks is used for placement of labor analgesia
  Epidural infusion: An epidural infusion will be started in both groups, regarding of the technique used for placement, and the same solution of Bupivacaine 0.0625% with 2mcg fentanyl/cc will be used in both groups
Period: Overall Study
Arm/Group | Ultrasound | No Ultrasound
Started | 12 | 20
Completed | 9 | 14
Not Completed | 3 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Data lost | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Ultrasound: Ultrasound guided CSE placed
  Ultrasound used for the correct interspace and midline position are identified for correct placement of the CSE analgesia.
  Epidural infusion - Bupivacaine 0.0625% with 2mcg fentanyl/cc
- No Ultrasound: CSE placed using palpation of anatomical landmarks
  No ultrasound: Palpation of anatomical landmarks is used for placement of labor analgesia
  Epidural infusion - Bupivacaine 0.0625% with 2mcg fentanyl/cc
- Total: Total of all reporting groups
Arm/Group | Ultrasound | No Ultrasound | Total
Number analyzed (Participants) | 9 | 14 | 23
Age, Customized [Count of Participants; unit: Participants]
  21 years and over | 9 | 14 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Learning Curve of Anesthesia Residents
Description: The success rate of epidural with each technique and improvement
Time Frame: 1 month
Population: Data not collected
Arm/Group | Ultrasound | No Ultrasound
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Attempts
Description: The number of attempts to locate the epidural space and midline position via ultrasound guided CSE technique.
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: attempts
Arm/Group | Ultrasound | No Ultrasound
Number analyzed (Participants) | 9 | 14
attempts | 1.333 [1 to 2] | 1.357 [1 to 3]

3. Secondary Outcome: Percentage of Accurate Epidural Placement
Description: Percentage of accurate epidural placement assessed by participant reporting pain 2 hours after CSE placed
Time Frame: 2 hours
Measure: Number; unit: percentage of accurate placement
Arm/Group | Ultrasound | No Ultrasound
Number analyzed (Participants) | 9 | 14
percentage of accurate placement | 66 | 86

4. Secondary Outcome: Number of Angle Adjustments in Space
Description: The number of angle adjustments of the epidural needle via ultrasound guided CSE technique.
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: adjustments
Arm/Group | Ultrasound | No Ultrasound
Number analyzed (Participants) | 9 | 14
adjustments | 1.78 [1 to 4] | 1.28 [1 to 4]

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Ultrasound | No Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-06-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02747238/Prot_001.pdf